CLINICAL TRIAL: NCT05868889
Title: Retrospective Multicenter Study of Elderly Patients With Ovarian Cancer Treated With Trabectedin and PLD According to SmPC
Brief Title: Retrospective Multicenter Study of Elderly Patients With Ovarian Cancer Treated With Trabectedin and PLD
Status: Completed | Type: Observational
Sponsor: Grupo Español de Investigación en Cáncer de Ovario (Other)
Responsible Party: Sponsor
Other Study IDs: GEICO 105-O
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Trabectedin; 1-dodecylpyridoxal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Trabectedin and PLD — The main treatment observed in this study is trabectedin in combination with PLD in elderly patients with platinum-sensitive relapsed ovarian cancer, according to the SmPC.

SUMMARY:
The median age at which ovarian cancer is diagnosed is 63 years (50-75). This is still a significant adverse factor for survival results. Seventy years can be considered the lower limit for the elderly term, since most of age-related changes occur later. Because of this, this group of patients is often not included in clinical trials and sometimes they do not receive adequate treatment. Little information is available on chemotherapy treatments in elderly patients. Data on the use of first-line chemotherapy in this population have recently been published. Trabectedin in combination with PLD is indicated for platinum-sensitive relapsed ovarian cancer and is an option for those patients in whom platinum is not the best option. There are some studies with trabectedin in combination with PLD in which some patients with this profile have been included, although not exclusively. Therefore, it is of interest to study the safety and efficacy profile of this treatment in elderly patients. With this information we will be able to know its real use in routine clinical practice at the national level in Spain in this population for which not much information is available. Safety and efficacy data (e.g. PFS, ORR, OS) will be collected retrospectively in order to draw conclusions about the combination of trabectedin + PLD, as a treatment option in this patient profile.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be signed by all patients participating in the study who can be interviewed in the hospital (accessible, alive patients) or absence of consent sheet must be signed by the investigator. Informed consent may not be required from unaccesible patients (dead, lost, etc.) according to ethics committee permissions and applicable law for retrospective studies in Spain.
* Adult women (≥70 years at the time of treatment initiation with trabectedin and PLD).
* Histological diagnosis of platinum-sensitive relapsed ovarian cancer (PFI ≥ 6 months).
* Treatment started with trabectedin and PLD (at least one cycle) as standard of care between January 1st 2015 and December 31st 2019.
* Patients must have received at least one cycle of trabectedin + PLD.

Exclusion Criteria:

* Patients without medical record available (lost, empty or unretrievable clinical information).
* Patients who explicitly refuse to participate in the study.

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adult women (≥ 70 years) diagnosed with platinum-sensitive relapsed ovarian cancer.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Serious and non-serious adverse events | 8 months
  Safety profile
Progression-free survival (PFS) | 8 months
  Time in months since first trabectedin + PLD dose date until radiological progression (or death due to any cause) according to RECIST 1.1 criteria
Overall response rate (ORR) | 8 months
  Number of patients having a best overall response (BOR) of complete response (CR) or partial response (PR), divided by the total number of response-evaluable patients (according to RECIST 1.1 criteria)
Disease control rate (DCR) | 8 months
  Percentage of patients having a complete response (CR), partial response (PR), or stable disease (SD) according to RECIST 1.1 criteria
Overall survival (OS) | 8 months
  Number of months since first trabectedin + PLD dose date until death due to any cause
Trabectedin + PLD treatment information (for both drugs) | 8 months
  Starting dose, total dose
Previous and subsequent treatments to trabectedin + PLD | 8 months
  Number of previous/subsequent treatments
Patient characteristics and medical history | 8 months
  Platinum-free interval (PFI)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT05868889/Prot_SAP_000.pdf